CLINICAL TRIAL: NCT05449951
Title: Effect of Dry Needling on Spasticity in Stroke Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Raheela IRB # 280-21
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Spastic Hemiplegia
Keywords: Dry needling; Modified Ashworth Scale; Goniometer; Range of Motion
MeSH Terms: conditions — Hemiplegia | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: There are two groups.Group A experimental group which receive dry needling protocol along with conventional therapy.Group B is control group which receive sustained stretching protocol along with conventional therapy.
Who Masked: Participant
Masking Description: The participants are blinded towards treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): This intervention was for three weeks in which there are 2 sessions per week. Sterile, disposable dry needles brand of JIAJAN with size of 0.30x40mm were used. Intervention was initiated after palpation of muscles(flexor carpi radials and flexor carpi ulnaris).First cleaning the area through alcohol swabs. There is a point for FCR in medial forearm, to that point 4 cm below and 1 cm medial to the midpoint of crease of elbow was needled. There is a point for FCU at the center of the proximal third segment of a line from the medial epicondyle to the ulnar styloid process was needled.Then, in swift in-and-out motions around 5mm vertical motions without rotation the needle was manipulated .About 1 minute Dry needling was executed for each targeted area, in respect to the patient's level of tolerance. This was monitored by the physiotherapist throughout the session by asking for regular verbal feedback
  Interventions: Other: Dry needling
- Sustained stretching (Other): The second group received sustained stretching protocol along with conventional therapy. Participants undergone the overall treatment sessions for three weeks (3weeks) and 2 sessions per week. The targeted muscles are wrist flexors (flexor carpi radials and flexor carpi ulnaris). Participants received 10 repetition with 30 seconds hold in each session for 10 minutes. Pre and post data in each session was measured through outcome measure tools
  Interventions: Other: sustained stretching

INTERVENTIONS:
Other: Dry needling — In dry needling filiform needle without a bore is used to mimic acupuncture t beyond the use of medicines. On the basis of purpose process and skill level it differs from acupuncture. DN is frequently used to treat pain caused by musculoskeletal structures, including as myofascial pain disorders
  Arms: Dry needling
Other: sustained stretching — sustained stretching is a treatment protocol in which muscle goes into a stretch position for period of time which reduce spasticity
  Arms: Sustained stretching

SUMMARY:
Stroke is a disruption of blood flow to brain either due to clot formation or rupturing of arteries.It is a leading cause of disability worldwide with many consequences and spasticity is one of them.Spasticity is a resistance to passive stretch which disturbs patient quality of life and interrupt activity of daily living.there are multiple options to treat spasticity which includes both pharmacological and non-pharmacological treatments.

DETAILED DESCRIPTION:
Stroke is a global issue and burden of disease is high in Asia.the burden of disease is alarming due to its consequences and spasticity is one of them.According to the lance definition clinical practice is still based which is too narrow. Spasticity, according to Lance, is a motor disease characterized by a velocity-dependent increase in tonic stretch reflexes (muscle tone) with excessive tendon jerks, due to hyper excitability stretch reflex.Furthermore, long-term untreated spasticity can cause discomfort, contractures, and deformities, which can lead to functional issues such as mobility limitations, reliance on (ADL), and a lower quality of life.There is multiple option to treat spasticity including pharmacological and rehabilitation Pharmacological treatments that can be focal or systematic and have partial effects and eventually need of physical therapy There are many PT procedures which includes stretching neurodevelopment techniques and many others to prevent spasticity.

ELIGIBILITY:
Inclusion Criteria:

- 1: Ischemic or hemorrhagic stroke and includes any of the artery 2: Hemiplegia 3: Chronic stroke (stroke at least 6 months before the trial) 4: Present a level of spasticity equal or greater than between 1 to 3 according to Modified Ashworth Scale.

5: Preserve cognitive capacity according to 6 cognitive items test (6CIT), Montreal cognitive assessment (MoCA) and Mini mental state examination (MMSE)

Exclusion Criteria:

1: Insurmountable fear of needles. 2: Wrist fracture. 3: Have received previous treatment with dry needling. 4: Have progressive or severe neurological disease.

-

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-08-04 (Estimated); Study Completion 2022-08-08 (Estimated)

PRIMARY OUTCOMES:
Modified Asworth sacle | 3 weeks
  it is used to measure spasticity which ranges from 0-4
Goniometer | 3 weeks
  to measure range of motion of wrist extensors of maximum range 70 degrees
Motor Assesment Scale | 3 weeks
  2 components of this scale is used to measure hand function recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Shifa tameer e millat university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuriakose D, Xiao Z. Pathophysiology and Treatment of Stroke: Present Status and Future Perspectives. Int J Mol Sci. 2020 Oct 15;21(20):7609. doi: 10.3390/ijms21207609. PMID 33076218
- [Background] Salom-Moreno J, Sanchez-Mila Z, Ortega-Santiago R, Palacios-Cena M, Truyol-Dominguez S, Fernandez-de-las-Penas C. Changes in spasticity, widespread pressure pain sensitivity, and baropodometry after the application of dry needling in patients who have had a stroke: a randomized controlled trial. J Manipulative Physiol Ther. 2014 Oct;37(8):569-79. doi: 10.1016/j.jmpt.2014.06.003. Epub 2014 Sep 8. PMID 25199825
- [Background] Hadi S, Khadijeh O, Hadian M, Niloofar AY, Olyaei G, Hossein B, Calvo S, Herrero P. The effect of dry needling on spasticity, gait and muscle architecture in patients with chronic stroke: A case series study. Top Stroke Rehabil. 2018 Jul;25(5):326-332. doi: 10.1080/10749357.2018.1460946. Epub 2018 Apr 23. PMID 29683410
- [Background] Ghaffari MS, Shariat A, Honarpishe R, Hakakzadeh A, Cleland JA, Haghighi S, Barghi TS. Concurrent Effects of Dry Needling and Electrical Stimulation in the Management of Upper Extremity Hemiparesis. J Acupunct Meridian Stud. 2019 Jun;12(3):90-94. doi: 10.1016/j.jams.2019.04.004. Epub 2019 Apr 23. PMID 31026521
- [Background] Sanchez-Mila Z, Salom-Moreno J, Fernandez-de-Las-Penas C. Effects of dry needling on post-stroke spasticity, motor function and stability limits: a randomised clinical trial. Acupunct Med. 2018 Dec;36(6):358-366. doi: 10.1136/acupmed-2017-011568. Epub 2018 Jul 9. PMID 29986902
- [Background] Hong CZ. Needling therapy for myofascial pain control. Evid Based Complement Alternat Med. 2013;2013:946597. doi: 10.1155/2013/946597. Epub 2013 Aug 26. No abstract available. PMID 24066015
- [Background] Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. Int J Sports Phys Ther. 2012 Jun;7(3):306-13. PMID 22666645